CLINICAL TRIAL: NCT04245722
Title: A Phase I, Open-Label, Multicenter Study of FT596 as a Monotherapy and in Combination With Rituximab or Obinutuzumab in Subjects With Relapsed/Refractory B-cell Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: FT596 as a Monotherapy and in Combination With Anti-CD20 Monoclonal Antibodies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT596-101
Record Dates: First submitted 2020-01-18; First posted 2020-01-29 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma, B-Cell; Chronic Lymphocytic Leukemia
Keywords: Lymphoma; Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Leukemia | interventions — Cyclophosphamide; fludarabine; Rituximab; obinutuzumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- FT596 Monotherapy, Lymphoma (Experimental): FT596 monotherapy in adult subjects with r/r B-cell Lymphoma
  Interventions: Drug: FT596; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT596 in Combination with Rituximab, Lymphoma (Experimental): FT596 in combination with Rituximab in adult subjects with r/r B-cell Lymphoma
  Interventions: Drug: FT596; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab; Drug: Bendamustine
- FT596 in Combination with Obinutuzumab, Lymphoma (Experimental): FT596 in combination with Obinutuzumab in adult subjects with r/r B-cell Lymphoma
  Interventions: Drug: FT596; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Obinutuzumab; Drug: Bendamustine
- FT596 Monotherapy, CLL (Experimental): FT596 monotherapy in adult subjects with r/r CLL
  Interventions: Drug: FT596; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT596 in Combination with Obinutuzumab, CLL (Experimental): FT596 in combination with Obinutuzumab in adult subjects with r/r CLL
  Interventions: Drug: FT596; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Obinutuzumab; Drug: Bendamustine

INTERVENTIONS:
Drug: FT596 — Experimental Interventional Therapy
Drug: Cyclophosphamide — Lympho-conditioning agent
Drug: Fludarabine — Lympho-conditioning agent
Drug: Rituximab — Monoclonal Antibody
  Other Names: Rituxan; Truxima; Ruxience
  Arms: FT596 in Combination with Rituximab, Lymphoma
Drug: Obinutuzumab — Monoclonal Antibody
  Other Names: Gazyva
  Arms: FT596 in Combination with Obinutuzumab, CLL; FT596 in Combination with Obinutuzumab, Lymphoma
Drug: Bendamustine — Conditioning agent
  Other Names: Bendeka; Treanda

SUMMARY:
This is a Phase I dose-finding study of FT596 as monotherapy and in combination with Rituximab or Obinutuzumab in subjects with relapsed/refractory B-cell Lymphoma or Chronic Lymphocytic Leukemia. The study will consist of a dose-escalation stage and an expansion stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

Diagnosis of B-cell lymphoma or CLL as described below:

B-Cell Lymphoma:

* Histologically documented lymphomas expected to express CD19 and CD20
* Relapsed/refractory disease following prior systemic immunochemotherapy regimen

Chronic Lymphocytic Leukemia (CLL):

* Diagnosis of CLL per iwCLL guidelines
* Relapsed/refractory disease following at least two prior systemic treatment regimens

ALL SUBJECTS:

* Capable of giving signed informed consent
* Age ≥ 18 years old
* Stated willingness to comply with study procedures and duration
* Contraceptive use for women and men as defined in the protocol

Key Exclusion Criteria:

ALL SUBJECTS:

* Females who are pregnant or breastfeeding
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥2
* Body weight <50 kg
* Evidence of insufficient organ function
* Receipt therapy within 2 weeks prior to Day 1 or five half-lives, whichever is shorter; or any investigational therapy within 28 days prior to Day 1
* Currently receiving or likely to require systemic immunosuppressive therapy
* Prior allogeneic hematopoietic stem cell transplant (HSCT) or allogeneic CAR-T within 6 months of Day 1, or ongoing requirement for systemic GvHD therapy
* Receipt of an allograft organ transplant
* Known active central nervous system (CNS) involvement by malignancy
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Clinically significant cardiovascular disease
* Known HIV infection
* Known active Hepatitis B (HBV) or Hepatitis C (HCV) infection
* Live vaccine <6 weeks prior to start of lympho-conditioning
* Known allergy to albumin (human) or DMSO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities within each dose level cohort | Day 29
Nature of dose-limiting toxicities within each dose level cohort | Day 29
Incidence, nature, and severity of adverse events (AEs) of FT596 as monotherapy and in combination with rituximab or obinutuzumab in r/r B-cell lymphomas and r/r chronic lymphocytic leukemia, with severity determined according to NCI CTCAE, v5.0 | Up to 15 years

SECONDARY OUTCOMES:
Investigator-assessed objective-response rate (ORR) | From baseline tumor assessment up to approximately 2 years after last dose of FT596
  Proportion of subjects who achieve a partial response (PR) or complete response (CR) per Lugano 2014 classification for lymphomas, a partial remission (PR) or complete remission (CR) per revised iwCLL guidelines for CLL.
Investigator-assessed duration of objective response (DOR) | Up to 15 years
  Defined as the duration from the first occurrence of a documented objective response (DOR) until the time of disease progression or relapse, or death from any cause, whichever occurs first, per Lugano 2014 classification for lymphomas or revised iwCLL guidelines for CLL.
Investigator-assessed duration of complete response (DoCR) | Up to 15 years
  Defined as the duration from the first occurrence of a documented complete response (CR) per Lugano 2014 classification for lymphomas or complete remission (CR) per revised iwCLL guidelines for CLL, until the time of disease progression or relapse, or death from any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 15 years
  Defined as the time from from first dose of lympho-conditioning to progressive disease (PD), or to the day of death for any reason, whichever occurs earlier, based on Lugano 2014 classification for lymphomas or revised iwCLL guidelines for CLL
Overall survival (OS), defined as the time from first dose of lympho-conditioning to death from any cause. | Up to 15 years
The pharmacokinetics of FT596 in peripheral blood will be reported as the relative percentage of product (FT596) DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points | Study Days: 1, 2, 4, 8, 11, 15, 18, 22, 29

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics
Locations (9):
- United States (9):
  - The University of Chicago, Chicago, Illinois
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute (Tennessee Oncology), Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - SCRI-TTI, San Antonio, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Hermanson DL, Moriarity BS, Kaufman DS. Human iPSC-Derived Natural Killer Cells Engineered with Chimeric Antigen Receptors Enhance Anti-tumor Activity. Cell Stem Cell. 2018 Aug 2;23(2):181-192.e5. doi: 10.1016/j.stem.2018.06.002. Epub 2018 Jun 28. PMID 30082067
- [Derived] Ghobadi A, Bachanova V, Patel K, Park JH, Flinn I, Riedell PA, Bachier C, Diefenbach CS, Wong C, Bickers C, Wong L, Patel D, Goodridge J, Denholt M, Valamehr B, Elstrom RL, Strati P. Induced pluripotent stem-cell-derived CD19-directed chimeric antigen receptor natural killer cells in B-cell lymphoma: a phase 1, first-in-human trial. Lancet. 2025 Jan 11;405(10473):127-136. doi: 10.1016/S0140-6736(24)02462-0. PMID 39798981